CLINICAL TRIAL: NCT03439059
Title: REducing SEDENTary Behaviour May Slow Cognitive Decline in Older Adults With Mild Cognitive Impairment: A Pilot Study
Acronym: RESEDENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESEDENT study
Record Dates: First submitted 2018-02-09; First posted 2018-02-20 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2019-01

CONDITIONS: Cognitive Impairment; Physical Functioning; Quality of Life
Keywords: Older adults; Sedentary behaviour; Assisted living; cognitive function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention- reducing SB (Experimental): prompted to do 10min of light physical activity 3x/day
  Interventions: Behavioral: Reducing Sedentary Behaviour Group
- Control (No Intervention): go about their normal daily living

INTERVENTIONS:
Behavioral: Reducing Sedentary Behaviour Group — Participants will be prompted to perform 10min of light physical activity (>1.5 METS) 3x/day for 6 weeks
  Arms: intervention- reducing SB

SUMMARY:
With the nation's fastest growing demographic being adults over 65, one in every three seniors is estimated to die from Alzheimer's Disease (AD). The strong correlation between AD and age, combined with the exponential growth of this demographic, highlights the need for non-pharmaceutical treatment/prevention strategies. Research has established a relationship between moderate to vigorous physical activity (PA) and improved cognitive functioning. However, there is insufficient evidence to support this relationship at the lower end of the PA spectrum. Assisted living facilities (ALF) are an easy target for reducing SB, as many individuals in these facilities have various functional limitations and therefore cannot meet the recommended PA guidelines. Older adults are also the most sedentary population, with results showing over 8.5+ hours daily spent in SB. ALF typically provide meals, laundry services as well as housekeeping duties, leaving the residents very susceptible to large amounts of SB. The primary purpose of my study is investigating how reducing sedentary behaviour (SB) in ALF will affect Alzheimer's Disease Assessment Scale-cognitive scores among older adults aged 65 and older with mild-to-moderate cognitive impairment. I will also investigate its effects on physical functioning with the Timed Up and Go test (TUG) and quality of life with the Short Form 36 (SF-36) Health Survey. Participants will be prompted to take a 10-minute light intensity PA break at three different time points throughout the day, reallocating SB to any task equating to over 1.5 metabolic equivalents. Positive findings may encourage ALF to implement policies and procedures regarding SB.

DETAILED DESCRIPTION:
Dementia is the leading cause of dependence and disability worldwide. With the nation's fastest growing demographic being adults over 65, the Lewy Body Dementia Association states that the current cost puts it higher than either heart disease or cancer; as the financial burden was estimated at $818 billion in 2015. Functional limitations such as a slower gait, muscle weakness (ex. grip strength), unintentional weight loss and self-reported exhaustion adds pressure on healthcare services. Older adults transitioning into assisted living facilities (ALF) will need assistance with activities of daily living; as this population is the most sedentary. Although exercise interventions show positive effects for the management of chronic diseases, as well as cognition and physical functioning, the Canadian Health Measures Survey reported that only 13% of older adults 60- 79 years old were meeting the physical activity (PA) guidelines set out by the World Health Organization. That said, research has yet to establish what benefits may come from the lower end of the PA spectrum; and there are no current guidelines for how long older adults should be sedentary. Research shows that large amounts of sedentary behaviour (SB) leads to an increased risk of all-cause mortality, independent from not meeting the PA guidelines (Ekelund et al., 2016). SB is defined as any waking behaviour characterized by an energy expenditure less than or equal to 1.5 metabolic equivalents while in a sitting or reclining posture. Alzheimer's Disease (AD) is the most common form of Dementia, accounting for 60-80% of cases; and Mild Cognitive Impairment (MCI) is generally used to refer to the transitional zone between normal cognitive functioning and clinically probable AD. With no current cure for AD, the need for effective non-pharmaceutical treatments are imperative.

The purpose of my study will be to investigate the effect of reducing SB on Alzheimer's Disease Assessment Scale-cognitive (ADAS-cog) scores among older adults aged 65 years and older with moderate cognitive impairment. Also, examine their changes in physical functioning and their quality of life. I hypothesize that the decline in ADAS-cog scores will be slower and physical scores as well as quality of life (QoL) scores will improve in the intervention group vs controls.

A clustered randomized control pilot study; involving an ALF in London, Ontario will be conducted. The intervention group will be prompted to take a 10-minute light intensity PA break three times throughout the day. The PA will be any task equating to over 1.5 metabolic equivalents and will be recorded in a simplified diary. Eligible subjects will undergo the following tests at baseline: 1) the Mini Mental State Examination and 2) the Community Healthy Activities Program for Seniors survey, 3) Timed Up and Go test (TUG) for physical functioning; 4) ADAS-cog for cognitive functioning; and 5) the Short Form- 36 Health Survey to assess QoL. Both groups will wear an activity tracker during a baseline period before the intervention to collect baseline levels of physical activity. Both groups will also be required to wear the activity monitor for a period during the intervention to check adherence. Following the intervention, the CHAMPS questionnaire will be re-administered along with the ADAS-cog, TUG and SF-36.

Research at the bottom end of the PA spectrum is crucial, as residents in ALF have various functional limitations; and many cannot meet the current PA guidelines. If improvements are shown from my study, this could contribute to the design of a policy that can be implemented into all ALF; lessening the burden on the health care system and loved ones.

ELIGIBILITY:
Inclusions:

* aged 65+ years old
* residing in the ALF permanently
* able to read, write and understand English
* answer "yes" to "do you have difficulty with your memory"
* get consent from their physician to participate in the study
* diagnosed with mild- moderate cognitive impairment by obtaining a score of 14-29, inclusive, on the Mini Mental State Examination (Folstein, Folstein, & McHugh, 1975).

Exclusions:

* any physical condition or disability disallowing participation in PA
* apparent evidence of any neurodegenerative disorders other than Alzheimer's disease
* score of 6 or higher on the Geriatric Depression Scale (Almeida, 1999), due to the apparent presence of clinically significant depressive symptoms and finally

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Alzheimers Disease Assessment Scale- Cognitive (ADAS-cog) | 10 weeks
  The ADAS-Cog Sub-Scale is the standard cognitive outcome measure used in clinical trials for patients with mild to moderate Alzheimer's disease. The test consists of 11 brief cognitive tests assessing memory, language, praxis, attention and other cognitive abilities. Scores range from 0 to 70, with higher scores indicating greater severity of cognitive impairment

SECONDARY OUTCOMES:
Short Form 36 Health Survey | 10 weeks
  Used for measuring functional health status and wellbeing in older adults. The questionnaire consists of 36 questions and is designed to measure eight multi-item dimensions, covering functional status, well being and overall evaluation of health.
Timed Up and Go test | 10 weeks
  A test for measuring basic functional mobility. It consists of the time taken (in seconds) to stand up from a standard arm chair, walk 3 m, turn around, and walk back to the chair and sit down again

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, Ph.D, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No